CLINICAL TRIAL: NCT03567720
Title: A Phase 2 Multi-Cohort, Open-Label Study of Intratumoral Tavokinogene Telseplasmid Plus Electroporation in Combination With Pembrolizumab +/- Chemotherapy in Patients With Inoperable Locally Advanced/Metastatic Triple-Negative Breast Cancer
Brief Title: Tavo and Pembrolizumab With or Without Chemotherapy in Patients With Inoperable Locally Advanced or Metastatic TNBC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: OncoSec Medical Incorporated (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OMS-I141 (KEYNOTE-890); KEYNOTE-890 (Other: Merck & Co); MK3475-890 (Other: Merck & Co)
Record Dates: First submitted 2018-06-13; First posted 2018-06-26 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Triple Negative Breast Cancer
Keywords: Metastatic; Inoperable Locally Advanced; TNBC; plasmid interleukin-12; tavokinogene telseplasmid; pembrolizumab; chemotherapy; pIL-12; Nab-paclitaxel; gemcitabine plus carboplatin; IL-12; IL12
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Neoplasm Metastasis | interventions — pembrolizumab; Taxes; Albumin-Bound Paclitaxel; Gemcitabine; Carboplatin

STUDY DESIGN:
Intervention Model Description: Phase 2, Multi-Cohort, Open-Label, Multi-Center Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- TAVO-EP plus IV pembrolizumab (Experimental): Intratumoral Tavokinogene Telseplasmid (tavo, pIL 12) plus Electroporation (ImmunoPulse) in Combination with Intravenous Pembrolizumab (Cohort enrollment completed)
  Interventions: Biological: tavokinogene telseplasmid; Biological: Pembrolizumab; Device: Immunopulse
- TAVO-EP plus IV pembrolizumab with chemotherapy (Experimental): Intratumoral Tavokinogene Telseplasmid (tavo, pIL 12) plus Electroporation (ImmunoPulse) in Combination with Intravenous Pembrolizumab along with treatment of an approved chemotherapy per standard of care (either nab-paclitaxel or gemcitabine plus carboplatin)
  Interventions: Biological: tavokinogene telseplasmid; Biological: Pembrolizumab; Device: Immunopulse; Drug: nab paclitaxel; Drug: gemcitabine plus carboplatin

INTERVENTIONS:
Biological: tavokinogene telseplasmid — Intratumoral tavokinogene telseplasmid delivered by electroporation every 6 weeks
  Other Names: pIL-12; tavo-EP
Biological: Pembrolizumab — Intravenous 3 weekly treatments
  Other Names: Keytruda
Device: Immunopulse — Device that administers electroporation
  Other Names: tavo-EP
Drug: nab paclitaxel — intravenous on days 1, 8 and 15 of each 28 day cycle
  Other Names: Abraxane
  Arms: TAVO-EP plus IV pembrolizumab with chemotherapy
Drug: gemcitabine plus carboplatin — intravenous on days 1 and 8 of every 21 days
  Other Names: Gemzar; Paraplatin
  Arms: TAVO-EP plus IV pembrolizumab with chemotherapy

SUMMARY:
This is a Phase 2, Multi-Cohort, Open-Label, Multi-Center Study. Cohort 1 will be a single-arm study of intratumoral tavokinogene telseplasmid (TAVO) plus electroporation (EP) in combination with pembrolizumab therapy. Cohort 2 will be a single-arm study of intratumoral TAVO-EP plus pembrolizumab along with treatment of an approved chemotherapy per standard of care (either nab-paclitaxel (Abraxane®) or gemcitabine (Gemzar®) plus carboplatin (Paraplatin®)) in participants with TNBC and no prior systemic therapy in the advanced or metastatic setting will be enrolled in this study.

DETAILED DESCRIPTION:
The study will include a screening period, treatment period (up to 2 years), a long-term follow-up period, and a survival follow-up period. Participants will be followed for disease status and survival for up to a total duration of 5 years from the time of first dose of study treatment.

Eligible subjects with accessible lesions will be treated with TAVO-EP on Days 1, 5 and 8 every 6 weeks for up to 18 weeks. Pembrolizumab IV will be administered at a dose of 200 mg on Day 1 every 3-weeks for up to 35 cycles (Q3W) or 400 mg on Day 1 every 6 weeks for up to 18 cycles (Q6W).

Eligible subjects will be enrolled in one of the following cohorts.

* Cohort 1 is a single-arm study of intratumoral TAVO-EP and pembrolizumab (Q3W) in participants with TNBC and at least 1 line of prior systemic therapy in the advanced or metastatic setting.
* Cohort 2 is a single-arm study of intratumoral TAVO-EP and pembrolizumab along with treatment with an approved chemotherapy per standard of care (either nab-paclitaxel (Abraxane®)or gemcitabine (Gemzar®) plus carboplatin (Paraplatin®)) in participants with TNBC and no prior systemic therapy in the advanced or metastatic setting. Participants enrolled on or after Protocol Version 7 will have baseline disease PD-L1 negative status defined as Dako 22C3 assay CPS <10.

For participants in Cohort 2 receiving nab-paclitaxel, the schedule for nab-paclitaxel is a separate 28-day cycle. The dosing regimen of nab-paclitaxel is 100 mg/m2 IV over 30 minutes on Days 1, 8, and 15 of each 28-day cycle.

For participants in Cohort 2 receiving gemcitabine plus carboplatin, the dosing regimen is gemcitabine 1000 mg/m² plus carboplatin area under the curve (AUC) 2 IV on Days 1 and 8 every 21 days.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with histologically confirmed diagnosis of inoperable locally advanced or metastatic TNBC.
2. The following prior cancer therapy requirements apply to specific cohorts:

   1. For Cohort 1 only, subjects must have received at least 1 prior line of systemic chemotherapy or immunotherapy that includes an approved regimen.
   2. For Cohort 2 only, subjects has had no prior systemic therapy in the advanced/metastatic setting and must not have progression or recurrence of disease within 6 months after the last dose of systemic neoadjuvant or adjuvant treatment, if applicable.
3. Subjects must have TNBC defined as estrogen (ER) receptor and progesterone (PR) receptor staining <10% and human epidermal growth factor receptor 2 (HER2) - negative defined as immunohistochemistry (IHC) 0 to 1+
4. For Cohort 2, the participant must meet each of the following criteria:

   1. Has baseline PD-L1 negative disease (defined as Dako 22C3 assay CPS<10 [or equivalent, per sponsor agreement]) with results provided prior to start of study drug dosing: Historic results or new local PD-L1 testing from tissue collected within 6 months and without intervening therapy prior to Cycle 1 Day 1
   2. Can provide a separate core or punch tumor biopsy collected at screening or archival tissue collected within 6 months (and without intervening therapy) prior to Cycle 1 Day 1
   3. Has at least one lesion suitable for biopsy on Cycle 2 Day 1 (preferably same lesion from which the screening sample was collected).
5. Subjects must not have disease that, in the opinion of the Investigator, is considered amenable to potentially curative treatment.
6. Age ≥ 18 years of age of day of signing informed consent.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
8. Life expectancy of at least 6 months.
9. Participant has measurable disease based on RECIST v1.1 and has at least one identified lesion (target or non-target) that is accessible (up to 1.5 cm from the skin surface) and in a safe location for intratumoral injection and electroporation.
10. Demonstrate adequate organ function. All screening laboratories should be performed within 10 days of treatment initiation.
11. Female participant of childbearing potential must have a negative pregnancy test (for serum or urine pregnancy test, within 72 hours or 24 hours, respectively, prior to receiving the first study drug administration). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
12. Female participant of childbearing potential must be willing to use an adequate method of contraception from the first day of study treatment (or 14 days prior to the initiation of study treatment for oral contraception) and through at least 120 days following the last day of study treatment.
13. Male participant is surgically sterile OR agrees to use an adequate method of contraception when having sex with women of childbearing potential and refrains from sperm donation during the study treatment period and at least 120 days following the last day of study treatment.
14. Participant is able and willing to give informed consent and to follow study instructions.

Exclusion Criteria:

1. Subject has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
2. Subject has a clinically active brain metastases or leptomeningeal metastases. Participant who has a previously treated brain metastases or untreated asymptomatic brain metastases ≤5 mm may participate provided that they are radiologically stable (ie, without evidence of progression based on imaging during study screening), clinically stable, and without requirement of steroid treatment for at least 14 days prior to the first dose of study treatment.
3. Subject has had an allogenic tissue/solid organ transplant.
4. Subjects with electronic pacemakers or defibrillators.
5. Subject who have a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
6. Subject has active hepatitis B (defined as HBsAg reactive) or active hepatitis C (defined as HCV RNA [qualitative] is detected). Note: Participant with a history of HBV or HCV controlled by ongoing viral suppression therapy is allowed.
7. Subject has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg/day of prednisone or equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
8. Subject has an active autoimmune disease that required systemic treatment in the past 2 years (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
9. Subject has received a live-virus or live-attenuated vaccine within 30 days prior to the first dose of study treatment. Note: Administration of killed vaccines are allowed.

   Seasonal flu vaccines and COVID-19 vaccines that do not contain live virus (including attenuated vaccines) are permitted.
10. Subject has severe hypersensitivity (≥Grade 3) to pembrolizumab or other anti-PD-1 monoclonal antibody therapy and/or any of its excipients.
11. For Cohort 2 only, participant has severe hypersensitivity (≥Grade 3) to or expected intolerance of the protocol-specified chemotherapy options. Participant must be able to tolerate at least one of the trial approved chemotherapy options.
12. Subject has received transfusion of blood products (including platelets or red blood cells) or colony stimulating factors (including G-CSF, GM-CSF, or recombinant erythropoietin) within 2 weeks prior to qualifying screening labs.
13. Subject has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
14. Subject has a history of interstitial lung disease.
15. Subject has an active infection requiring systemic therapy.
16. Subject has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.
17. Participant has not recovered (ie, ≤Grade 1 or at baseline) from adverse events (AEs) due to a previously administered agent.
18. Subject has received any systemic anti-cancer agent or other local anti-cancer immunotherapy within 14 days prior to the start of study treatment.
19. Subject has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
20. Subject is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2018-10-11 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Objective Response Rate (ORR) | Approximately 2 years
  ORR by Investigator review based on RECIST v1.1
Cohort 2: Objective Response Rate (ORR) | Approximately 2 years
  ORR by Investigator review based on RECIST v1.1

SECONDARY OUTCOMES:
Duration of Response (DOR) | Approximately 2 years
  Cohort 1 & Cohort 2: DOR by Investigator based on RECIST v1.1
Progression Free Survival (PFS) | Approximately 2 years
  Cohort 1 & Cohort 2: PFS by Investigator based on RECIST v1.1
Immune Progression Free Survival (iPFS) | Approximately 2 years
  Cohort 1 & Cohort 2: iPFS by Investigator review based on iRECIST
Immune Objective Response Rate (iORR) | Approximately 2 years
  Cohort 1 & Cohort 2: iORR by Investigator review based on iRECIST
Disease Control Rate (DCR) | Approximately 2 years
  Cohort 1 & Cohort 2: DCR by Investigator based on RECIST v1.1
Overall Survival | Approximately 2 years
  Cohorts 1 and 2: Overall Survival for Cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Bridget O'Keeffe, Study Director — OncoSec Medical Incorporated
Locations (14):
- United States (10):
  - University of Arizona, Tucson, Arizona
  - UC San Diego, La Jolla, California
  - Stanford University Medical Center, Palo Alto, California
  - The Lundquist Institute, Torrance, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - Virginia Cancer Specialists, Fairfax, Virginia
  - University of Washington, Seattle Cancer Care Alliance, Seattle, Washington
- Australia (4):
  - Westmead Hospital, Westmead, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Calvary Central Districts Hospital, Elizabeth Vale, South Australia
  - Box Hill Hospital, Box Hill, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jacobs L, Yshii L, Junius S, Geukens N, Liston A, Hollevoet K, Declerck P. Intratumoral DNA-based delivery of checkpoint-inhibiting antibodies and interleukin 12 triggers T cell infiltration and anti-tumor response. Cancer Gene Ther. 2022 Jul;29(7):984-992. doi: 10.1038/s41417-021-00403-8. Epub 2021 Nov 9. PMID 34754076